CLINICAL TRIAL: NCT03518957
Title: A Randomized Controlled Study of a 12-week Exercise Intervention Program Versus Observation in Early Stage Breast Cancer Patients on the Impact on Mental Health, Quality of Life and Immune Markers
Brief Title: 12-week Exercise Intervention Program Versus Observation in Early Stage Breast Cancer Patients on the Impact on Mental Health, Quality of Life and Immune Markers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/01283
Record Dates: First submitted 2018-03-27; First posted 2018-05-08 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention (Experimental): Patients who are randomised to this arm will be enrolled to the exercise programme.
  Interventions: Behavioral: Exercise
- Non-exercise (No Intervention): Patients who are randomised to the non-exercise group can continue their daily and physical activities as they normally would.

INTERVENTIONS:
Behavioral: Exercise — Week 1: Patients will undergo an introductory session where the occupational therapist will assess the general condition and physical fitness of the subjects.
  Week 1 to Week 12: Group exercise sessions supervised by a physiotherapist, twice per week, each session lasting 1 hour, with no more than 8 participants in each group exercise session. The exercise regimen for each session will be personally tailored for the subjects, and will include stretching, cardiovascular and strength training, and cooling down exercises.
  Week 12 onwards: Patients will receive phone calls- monthly for the first 6 months and then 3 monthly up to the 2-year mark, to encourage them to continue with their exercise regimen at home.
  Arms: Exercise intervention

SUMMARY:
Exercise in early breast cancer patients has the potential to improve depression, anxiety, fatigue, quality of life and even survival. The effects of exercise may come about by way of changes in weight, immune markers and telomere length, but data on this so far has not been conclusive. To better understand the physical, psychological, and biological effects of exercise on breast cancer survivorship, the investigators propose to perform a phase III randomized controlled trial of a 12-week exercise intervention program versus usual care in early stage breast cancer patients, and will follow up the patients prospectively for 5 years, with serial assessment of physical and functional activity, QoL, depression and anxiety scores, telomere length and plasma immune markers.

DETAILED DESCRIPTION:
In this study, 304 eligible patients will be randomized 1:1 to a 12-week exercise intervention program versus observation, and stratified by two factors: received adjuvant chemotherapy versus not, and age<50 versus age ≥50 years.

Breast cancer and its treatment can have both physical and psychological sequelae, which can persist many years after diagnosis. Physical effects include higher rates of pain, fatigue and decline in physical function, while psychological effects include depression and anxiety. In particular, depression spectrum syndromes occur in 20-50% of people with cancer, and in 1.5-46% of people with breast cancer. In a recent study conducted locally at the National University Cancer Institute, Singapore (NCIS), it was found that 27% of newly diagnosed cancer patients have caseness for depression and 44% have caseness for anxiety, as measured using the Hospital Anxiety and Depression scale. Breast cancer is also associated with weight gain - as many as 50-96% of women, especially those undergoing chemotherapy, experience sarcopenic weight gain during treatment, in the range of 2.5-6.2kg. Patients do not tend to return to their pre-diagnosis weight. With respect to quality of life (QoL), poorer QoL occurs in the short term, whereas long-term survivors tend to have a good overall QoL, albeit with an increase in some specific problems like lymphoedema and sexual dysfunction. Some of these measures predict overall survival and risk of recurrence - low levels of psychological distress and low fatigue independently predicted longer recurrence-free and overall survival, and lack of anxiety predicted longer recurrence-free survival. Obesity is also a poor prognostic factor and increases the risk of recurrence.

Telomere length (TL), which generally shortens with ageing, may also be implicated - in a study of breast cancer patients with or without insomnia, those with insomnia were reported to have higher rates of depression, fatigue and anxiety, and shorter TLs. Furthermore, breast cancer patients who were engaged in at least moderate physical activity had significantly longer TLs than those who did not, although there was no correlation between depression and shorter TLs in this study.Another study in prostate cancer patients showed that 3 months of comprehensive lifestyle changes after diagnosis was associated with increased telomere lengths and reduced telomerase activity after 5 years of follow-up.

To better understand the physical, psychological, and biological effects of exercise on breast cancer survivorship, the investigators propose to perform a phase III randomized controlled trial of a 12-week exercise intervention program versus usual care in early stage breast cancer patients, and will follow up the patients prospectively for 5 years, with serial assessment of physical and functional activity, QoL, depression and anxiety scores, telomere length and plasma immune markers.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 21-70 years
* Histological or cytological diagnosis of breast carcinoma
* Stage I-III breast cancer
* Has undergone curative breast cancer surgery with no clinically measurable tumor
* Between 4-12 weeks from the last adjuvant radiotherapy or chemotherapy session, if given, whichever is later. Patients who do not receive adjuvant chemotherapy or radiotherapy can be enrolled and will be randomized within 4-12 weeks of breast cancer surgery.
* Able to sign informed consent
* Able to adhere to study procedures

Exclusion Criteria:

* Cardiovascular, respiratory, or musculoskeletal problems that preclude moderate physical activity
* Major medical problems deemed by the investigator to be unsuitable for enrollment

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females will be included, as this is a study on breast cancer
Enrollment: 304 (Estimated)
Dates: Start 2015-03-12 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Improved mental health | 12 months
  Based on the HADS (Hospital Anxiety and Depression Scale) questionnaire, we define a score of ≥8/21 as caseness for anxiety or depression

SECONDARY OUTCOMES:
Adherence rate | 16 weeks
  Subjects are considered to have adhered to the 12-week exercise regimen if they have completed at least 20 scheduled sessions over a period of no longer than 16 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carayol M, Bernard P, Boiche J, Riou F, Mercier B, Cousson-Gelie F, Romain AJ, Delpierre C, Ninot G. Psychological effect of exercise in women with breast cancer receiving adjuvant therapy: what is the optimal dose needed? Ann Oncol. 2013 Feb;24(2):291-300. doi: 10.1093/annonc/mds342. Epub 2012 Oct 5. PMID 23041586
- [Background] Kolden GG, Strauman TJ, Ward A, Kuta J, Woods TE, Schneider KL, Heerey E, Sanborn L, Burt C, Millbrandt L, Kalin NH, Stewart JA, Mullen B. A pilot study of group exercise training (GET) for women with primary breast cancer: feasibility and health benefits. Psychooncology. 2002 Sep-Oct;11(5):447-56. doi: 10.1002/pon.591. PMID 12228878